CLINICAL TRIAL: NCT00734487
Title: Age-Related Eye Disease Study 2 Ancillary Spectral Domain Optical Coherence Tomography Study
Brief Title: AREDS 2 Ancillary Spectral Domain Optical Coherence Tomography Study
Acronym: A2ASDOCT
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00001749; Genentech FVF4400
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Age Related Macular Degeneration
Keywords: Spectral Domain Optical Coherence Tomography; Optical Coherence Tomography; AREDS2; AMD; Age-related macular degeneration; Drusen
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. AREDS2 subjects: Subjects enrolled in the AREDS2 clinical trial with a diagnosis of age-related macular degeneration.
- 2. Controls: Age-matched subjects without retinal pathology

SUMMARY:
The purpose of this study is to identify whether changes in age-related macular degeneration (AMD) over time as seen with spectral domain optical coherence tomography (SDOCT) imaging, can be used to predict vision loss and the advancement of AMD in people at moderate to high risk for progression.

DETAILED DESCRIPTION:
The primary objective of this study is to identify whether SDOCT patterns such as: drusen size, OCT reflectivity within drusen, photoreceptor (PR)change over drusen, microfoci of subretinal fluid (SRF), or retinal thickening are predictive of vision loss, progression of drusen, progression of photoreceptor loss over drusen, development of choroidal neovascularization (CNV), or development of geographic atrophy (GA).

The secondary objectives of this study are:

1. To define the relationship between SDOCT imaging, autofluorescence (AF)imaging, and color photographic or other fundus imaging of AREDS 2 patients in both a cross-sectional study of baseline data and a longitudinal study in data collected over the 5 year AREDS 2 study.
2. To compare the extent of geographic atrophy on SDOCT versus color photographs and autofluorescence.
3. To evaluate whether the SDOCT outcome measures differ significantly between AREDS 2 patients randomized to different oral supplements in the AREDS2.

ELIGIBILITY:
Inclusion Criteria:

AMD subjects and controls

* Men and women between the ages of 50 and 85 years

AMD subjects

* Enrollment in the AREDS 2 trial;
* Macular status ranges from large drusen in both eyes or large drusen in one eye and advanced AMD (neovascular AMD or geographic atrophy) in the fellow eye

Exclusion Criteria:

* Ocular media not clear enough to allow good fundus photography.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The A2A SDOCT study will recruit AMD subjects from the AREDS 2 study population at 4 AREDS 2 Study Centers. Controls will be recruited from Duke University Eye Center and Emory University.
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2008-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures are the percent of eyes developing CNV, mean change in visual acuity, and change in drusen volume, area of GA and photoreceptor layer thickness from SDOCT centered on the fovea. | 2 years and 5 years

SECONDARY OUTCOMES:
Drusen area measured from SDOCT versus from color fundus photographs. Mean change in drusen area reproducibility of measurements using these techniques. | 2 years and 5 years
Grading of drusen type, presence or absence of fluid, photoreceptor loss or retinal thickening from SDOCT versus from color fundus photographs at each timepoint. | 2 years and 5 years
Correlation between SDOCT imaging and autofluorescence imaging and onset of geographic atrophy. | 2 years and 5 years
Measurement of area of GA from SDOCT images versus color fundus photos versus AF images. | 2 years and 5 years
To evaluate whether the SDOCT outcome measures differ significantly between AREDS 2 patients randomized to different oral supplements in the AREDS2. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Toth, MD, Study Chair — Duke Health; Thomas Hwang, MD, Principal Investigator — Devers Eye Institute; Baker Hubbard, MD, Principal Investigator — Emory University Eye Center; Wai T Wong, MD, PhD, Principal Investigator — National Eye Institute (NEI)
Locations (4):
- United States (4):
  - Emory University Eye Center, Atlanta, Georgia
  - National Eye Institute, Bethesda, Maryland
  - Duke University Eye Center, Durham, North Carolina
  - Devers Eye Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
All findings resulting from the A2A SDOCT study will be prepared for publication in peer-reviewed journals and posted on PubMed Central once accepted.
  We are supportive of efforts by publishers and professional societies to develop technologies for on-line publishing of entire experimental datasets. We will archive experimental results and findings from the proposed project for at least the duration of the project, and make the underlying datasets available to other researchers upon request.

REFERENCES:
- [Background] Folgar FA, Yuan EL, Sevilla MB, Chiu SJ, Farsiu S, Chew EY, Toth CA; Age Related Eye Disease Study 2 Ancillary Spectral-Domain Optical Coherence Tomography Study Group. Drusen Volume and Retinal Pigment Epithelium Abnormal Thinning Volume Predict 2-Year Progression of Age-Related Macular Degeneration. Ophthalmology. 2016 Jan;123(1):39-50.e1. doi: 10.1016/j.ophtha.2015.09.016. Epub 2015 Nov 12. PMID 26578448
- [Background] Farsiu S, Chiu SJ, O'Connell RV, Folgar FA, Yuan E, Izatt JA, Toth CA; Age-Related Eye Disease Study 2 Ancillary Spectral Domain Optical Coherence Tomography Study Group. Quantitative classification of eyes with and without intermediate age-related macular degeneration using optical coherence tomography. Ophthalmology. 2014 Jan;121(1):162-172. doi: 10.1016/j.ophtha.2013.07.013. Epub 2013 Aug 29. PMID 23993787
- [Background] Folgar FA, Chow JH, Farsiu S, Wong WT, Schuman SG, O'Connell RV, Winter KP, Chew EY, Hwang TS, Srivastava SK, Harrington MW, Clemons TE, Toth CA. Spatial correlation between hyperpigmentary changes on color fundus photography and hyperreflective foci on SDOCT in intermediate AMD. Invest Ophthalmol Vis Sci. 2012 Jul 9;53(8):4626-33. doi: 10.1167/iovs.12-9813. PMID 22589439
- [Background] Chiu SJ, Izatt JA, O'Connell RV, Winter KP, Toth CA, Farsiu S. Validated automatic segmentation of AMD pathology including drusen and geographic atrophy in SD-OCT images. Invest Ophthalmol Vis Sci. 2012 Jan 5;53(1):53-61. doi: 10.1167/iovs.11-7640. PMID 22039246
- [Background] Yiu G, Pecen P, Sarin N, Chiu SJ, Farsiu S, Mruthyunjaya P, Toth CA. Characterization of the choroid-scleral junction and suprachoroidal layer in healthy individuals on enhanced-depth imaging optical coherence tomography. JAMA Ophthalmol. 2014 Feb;132(2):174-81. doi: 10.1001/jamaophthalmol.2013.7288. PMID 24336985
- [Background] Yiu G, Chiu SJ, Petrou PA, Stinnett S, Sarin N, Farsiu S, Chew EY, Wong WT, Toth CA. Relationship of central choroidal thickness with age-related macular degeneration status. Am J Ophthalmol. 2015 Apr;159(4):617-26. doi: 10.1016/j.ajo.2014.12.010. Epub 2014 Dec 17. PMID 25526948
- [Background] Christenbury JG, Folgar FA, O'Connell RV, Chiu SJ, Farsiu S, Toth CA; Age-related Eye Disease Study 2 Ancillary Spectral Domain Optical Coherence Tomography Study Group. Progression of intermediate age-related macular degeneration with proliferation and inner retinal migration of hyperreflective foci. Ophthalmology. 2013 May;120(5):1038-45. doi: 10.1016/j.ophtha.2012.10.018. Epub 2013 Jan 23. PMID 23352193
- [Background] Leuschen JN, Schuman SG, Winter KP, McCall MN, Wong WT, Chew EY, Hwang T, Srivastava S, Sarin N, Clemons T, Harrington M, Toth CA. Spectral-domain optical coherence tomography characteristics of intermediate age-related macular degeneration. Ophthalmology. 2013 Jan;120(1):140-50. doi: 10.1016/j.ophtha.2012.07.004. Epub 2012 Sep 8. PMID 22968145
- [Background] Chiu SJ, Li XT, Nicholas P, Toth CA, Izatt JA, Farsiu S. Automatic segmentation of seven retinal layers in SDOCT images congruent with expert manual segmentation. Opt Express. 2010 Aug 30;18(18):19413-28. doi: 10.1364/OE.18.019413. PMID 20940837
- [Background] Jain N, Farsiu S, Khanifar AA, Bearelly S, Smith RT, Izatt JA, Toth CA. Quantitative comparison of drusen segmented on SD-OCT versus drusen delineated on color fundus photographs. Invest Ophthalmol Vis Sci. 2010 Oct;51(10):4875-83. doi: 10.1167/iovs.09-4962. Epub 2010 Apr 14. PMID 20393117
- [Background] Veerappan M, El-Hage-Sleiman AM, Tai V, Chiu SJ, Winter KP, Stinnett SS, Hwang TS, Hubbard GB 3rd, Michelson M, Gunther R, Wong WT, Chew EY, Toth CA; Age-related Eye Disease Study 2 Ancillary Spectral Domain Optical Coherence Tomography Study Group. Optical Coherence Tomography Reflective Drusen Substructures Predict Progression to Geographic Atrophy in Age-related Macular Degeneration. Ophthalmology. 2016 Dec;123(12):2554-2570. doi: 10.1016/j.ophtha.2016.08.047. Epub 2016 Oct 25. PMID 27793356
- [Background] Sleiman K, Veerappan M, Winter KP, McCall MN, Yiu G, Farsiu S, Chew EY, Clemons T, Toth CA; Age-Related Eye Disease Study 2 Ancillary Spectral Domain Optical Coherence Tomography Study Group. Optical Coherence Tomography Predictors of Risk for Progression to Non-Neovascular Atrophic Age-Related Macular Degeneration. Ophthalmology. 2017 Dec;124(12):1764-1777. doi: 10.1016/j.ophtha.2017.06.032. Epub 2017 Aug 26. PMID 28847641
- See also: Age-Related Eye Disease Study 2 — http://www.areds2.org
- See also: Age-Related Eye Disease Study 2 (AREDS2) registry at ClinicalTrials.gov — http://clinicaltrials.gov/ct2/show/NCT00345176?term=AREDS2&rank=1